CLINICAL TRIAL: NCT07371897
Title: A Randomized, Open-label, Multi-center Phase III Clinical Study of Toripalimab Combined With Cisplatin and Docetaxel Versus Toripalimab Alone as Neoadjuvant Therapy for Locally Advanced Head and Neck Squamous Cell Carcinoma
Brief Title: Toripalimab ± Chemo as Neoadjuvant Therapy in LA-HNSCC: A Phase III Trial
Acronym: SHINE
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Xuekui Liu, Chief Physician, Department of Head and Neck Surgery, Sun Yat-sen University Cancer Center; Principal Investigator of the SHINE Study, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYSUCC-HN-2024-SHINE
Record Dates: First submitted 2026-01-19; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Head and Neck Squamous Cell Carcinoma HNSCC
Keywords: Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Docetaxel; Cisplatin; toripalimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Toripalimab monotherapy (Experimental): Participants receive two 3-week cycles of toripalimab 240 mg IV before undergoing radical surgery, followed by post-operative radiotherapy or chemoradiotherapy plus 12 additional cycles of toripalimab.
  Interventions: Drug: Toripalimab
- Toripalimab + chemotherapy (Experimental): Participants receive two 3-week cycles of toripalimab 240 mg IV combined with docetaxel 75 mg/m² and cisplatin 75 mg/m² before radical surgery, followed by post-operative radiotherapy or chemoradiotherapy plus 12 additional cycles of toripalimab.
  Interventions: Drug: Docetaxel and Cisplatin; Drug: Toripalimab

INTERVENTIONS:
Drug: Docetaxel and Cisplatin — Neoadjuvant chemotherapy: docetaxel 75 mg/m² IV Day 1 + cisplatin 75 mg/m² IV Day 1, repeated every 21 days for 2 cycles, given together with toripalimab in the combination arm.
  Other Names: Taxotere；Platinol
  Arms: Toripalimab + chemotherapy
Drug: Toripalimab — Humanised anti-PD-1 IgG4κ monoclonal antibody. 240 mg IV infusion Day 1 of each 21-day cycle for 2 neoadjuvant cycles, then 3 cycles concurrent with post-op radiotherapy/chemoradiotherapy, followed by 12 adjuvant cycles every 3 weeks.

SUMMARY:
This study compares two short pre-surgery treatments for locally advanced head and neck squamous cell cancer to see which one keeps the cancer from coming back longer.

Eligible patients (18-70 years, newly diagnosed, operable) will be randomly assigned to receive either toripalimab (immunotherapy) alone or toripalimab plus two cycles of chemotherapy (docetaxel and cisplatin). After the two cycles, all patients will have standard surgery followed by radiation (or chemo-radiation).

We will track tumor response, side effects, and quality of life. Possible benefits: tumor shrinkage and lower chance of recurrence; possible risks: low blood counts, rash, tiredness, or other drug-related side effects.

Taking part is voluntary and you can leave the study at any time.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed, newly diagnosed, non-metastatic, operable locally advanced head-and-neck squamous cell carcinoma (oral cavity, larynx, hypopharynx, or oropharynx) Stage III-IVA (p16-positive oropharynx T4N0-N2; p16-negative oropharynx III-IVA; larynx/hypopharynx/oral cavity III-IVA) PD-L1 CPS ≥ 1 Age 18-70 years ECOG performance status 0-1 Adequate organ function (ANC ≥ 2.0×10⁹/L, platelets ≥ 100×10⁹/L, TBIL < 1.5×ULN, ALT/AST < 1.5×ULN, creatinine < 1.5×ULN) No prior head-and-neck cancer surgery or radiotherapy No other malignancy within 5 years Signed informed consent

Exclusion Criteria:

* Previous systemic anti-cancer therapy for head-and-neck cancer Known hypersensitivity to study drugs Active or untreated hepatitis B/C, HIV positivity Severe cardiac, pulmonary, liver, or renal insufficiency precluding surgery Pregnancy or lactation Psychiatric or social conditions preventing compliance Organ transplant on chronic immunosuppression

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Estimated)
Dates: Start 2026-06-30 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
2-year Event-Free Survival | From randomisation to 24 months
  Proportion of patients alive and free from locoregional recurrence, distant metastasis, second primary tumor, or death from any cause within 24 months after randomisation, assessed per modified RECIST 1.1.
2-year Event-Free Survival (EFS) | From randomisation to 24 months
  Proportion of patients alive and free from locoregional recurrence, distant metastasis, second primary tumor, or death from any cause within 24 months after randomisation, assessed per modified RECIST 1.1.

IPD SHARING:
Plan to Share IPD: Undecided